CLINICAL TRIAL: NCT00005581
Title: Epirubicin Plus Paclitaxel Versus Cyclophosphamide, Epirubicin and 5-Fluorouracil as Adjuvant Treatment of Node Positive Breast Cancer Patients: A Controlled Randomized Phase III Study
Brief Title: Combination Chemotherapy in Treating Women With Stage II or Stage III Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067266; INRC-GONO-MIG-5; NCI-V99-1562
Record Dates: First submitted 2000-05-02; First posted 2004-05-20 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Fluorouracil; Paclitaxel

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of chemotherapy is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of combination chemotherapy in treating women who have stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall survival and disease free survival after adjuvant chemotherapy with epirubicin plus paclitaxel versus cyclophosphamide, epirubicin, and fluorouracil in women with stage IIA, IIB, or III breast cancer. II. Compare quality of life in these women with these treatment regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms within 35 days of surgery. Arm I: Patients receive epirubicin IV followed by paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for 4 courses. Arm II: Patients receive cyclophosphamide IV, epirubicin IV, and fluorouracil IV on day 1. Treatment repeats every 21 days for 6 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who are postmenopausal, or premenopausal and hormone receptor positive, receive tamoxifen orally once a day for 5 years starting on day 1. Patients receive radiotherapy to residual breast after 4 courses of chemotherapy. Quality of life is assessed. Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 1,000 patients will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIA, IIB, or III breast cancer treated with radical surgery (e.g., mastectomy, quadrantectomy, tumorectomy) and axillary lymph node dissection Positive axillary lymph nodes No more than 9 metastatic lymph nodes No distant metastases or local or locoregional disease No more than 5 weeks between surgery and beginning of study Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 70 and under Sex: Female Menopausal status: Not specified Performance status: ECOG 0 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Transaminases, alkaline phosphatase, and gamma glutamyltransferase no greater than 1.5 times upper limit of normal Renal: Not specified Cardiovascular: No heart disease that precludes use of anthracyclines (i.e., myocardial infarction, uncontrolled angina pectoris, uncontrolled arrhythmias, or valve disease) Other: No concurrent pathology that precludes use of antineoplastic drugs No mental retardation or psychiatric disease that precludes study No other current or prior malignancy within the past 10 years except squamous or basal cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No prior antineoplastic hormonal therapy Radiotherapy: No postoperative radiotherapy except to residual breast Surgery: See Disease Characteristics

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Rosso, MD, Study Chair — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (25):
- Italy (25):
  - Ospedale San Lazzaro, Alba
  - Ospedale Civile di Asti, Asti
  - Ospedale Oncologico A. Businco, Cagliari
  - Santo Spirito Hospital, Casale Monferato
  - Ospedale Santa Croce, Cuneo
  - Ospedale Galliera Oncologia, Genoa
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospendale S. Andrea EST, La Spezia
  - Ospedale Civile di Livorno, Livorno
  - Carlo Poma Hospital, Mantova
  - Azienda USSL NO 8, Merate
  - Instituto Scientifico H.S. Raffaele, Milan
  - Ospedale Santa Croce, Moncalieri
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale St. Santa Chiara, Pisa
  - USL NO 1, Sanremo
  - Azienda U.S.L. 1 - Sassari, Sassari
  - Ospedale S. Paolo, Savona
  - Osp. Civile USL 18, Sestri Lev.
  - Ospedale Sant Anna, Torino
  - Ospedale Evangelico Valdese, Torino
  - OIRM - Sant Anna, Torino
  - Ospedale Mauriziano Umberto I, Torino
  - Ospedale Maggiore dell' Universita, Trieste
  - Ospedale Molinette, Turin